CLINICAL TRIAL: NCT03590483
Title: Maternal and Perinatal Outcomes in Spontaneous Twins Versus Twins Conceived by Ovulation Induction and Assisted Reproductive Techniques: A Cross Section Study Within One Year
Brief Title: Outcomes in Spontaneous and ART Twin Pregnancies
Status: Completed | Type: Observational
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Shahla Alalaf, professor, Hawler Medical University
Other Study IDs: SAlalaf
Record Dates: First submitted 2018-06-16; First posted 2018-07-18 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Neonatal SEPSIS; Perinatal Mortality; Maternal Morbidity
Keywords: Twins; ART; Induction of Ovulation; Perinatal mortality
MeSH Terms: conditions — Neonatal Sepsis; Perinatal Death

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During the last decades, assisted reproductive technique has been transformed from a miracle to real and has become widely used for treatment human infertility.

this was associated with increased the rate of twin pregnancies

DETAILED DESCRIPTION:
Twin pregnancies are associated with an increased risk of maternal mortality & morbidity and an increase in the incidence of neonatal morbidity and mortality compared to singleton pregnancy.

The heterogeneous results reported so far can also depend on differences in the studied populations and/or in the management approach to twin pregnancy, variability in data regarding neonatal and maternal outcomes.

Evidence on pregnancy outcomes of twins conceived by artificial reproductive technology (ART) compared with those naturally conceived (NC) is conflicting, A 2004 systematic review and a large 2008 study both were praised that in cases of twin pregnancy after assisted conception the perinatal mortality is significantly lower, when compared with those spontaneously conceived .

ELIGIBILITY:
Inclusion Criteria:

* Twin delivered >24-week gestational age
* weight ≥ 500g
* Diachronic diamniotic twins.

Exclusion Criteria:

* Intrauterine fetal deaths
* Higher-order multiple pregnancies
* Deliveries complicated by early vanishing fetuses
* Twin pregnancies reduced to singleton
* Triple pregnancy reduced to twin.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Twin delivery was identified when coming to outpatient clinic & labour ward into two groups, first group iatrogenic conceived twins (either ART, or medical ovulation induction mainly clomiphene citrate and gonadotrophins).The second group is a twin pregnancy who conceived naturally .
  Demographic characters, maternal and neonatal outcomes were compared in both groups
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Maternal diabetes using glucose tolerance test | up to 7 days postpartum
  The diagnosis of GDM was based a fasting plasma glucose level of ≥5.6 mmol/L with 2 h plasma glucose level of ≥7.8 mmol/L
Hypertension during pregnancy and preeclampsia diagnosed using ACOG guideline a) weight in kilogram b) Apgar score in first and 10th minutes c)Admission to neonatal intensive acre unit measured in days | up to 1 week postpartum
  Systolic and diastolic blood pressure equal or more than140/90 mm Hg measured on two or more occasions after 20 weeks of gestation in previously normotensive women, with or without proteinuria (proteinuria of >100 mg/dL by urine analysis, or >300 mg/24 h)
Maternal anemia using WHO criteria | up to 1 week
  Hemoglobin level less than 11gm/dl
Postpartum hemorrhage | up to 1 week
  Bleeding from genital tract of 500 mL or more vaginally
Neonatal weight in kilogram | up to 7 days
  categorized as extreme low birth weight (LBW) for <1000 g, very LBW for 1000-1500 g, LBW for 1500-2500 g, and normal birth weight for >2500 g
Neonatal Apgar(Appearance, Pulse, Grimace, Activity, and Respiration) score | first and fifth minute of life
  Apgar scores includes 10 sores , 2 for each . The Apgar score was classified as severely depressed <0-3>, moderately depressed<4-6> and excellent condition<7-10>
Admission to neonatal care unit in days | up to 7 days
  Fetal care unit

SECONDARY OUTCOMES:
Maternal mode of delivery | during labor
  Cesarean section or vaginal delivery

CONTACTS AND LOCATIONS:
Overall Officials: Diana Y. Rashid, Principal Investigator — Maternity Teaching Hospital; Shahla K. Alalaf, Study Director — Hawler Medical University, College of Medicine
Locations (1):
- Kurdistan Board for Medical speciality, Erbil, Kurdistan Region, Iraq